CLINICAL TRIAL: NCT05999968
Title: A Phase 1b Study of Abemaciclib Plus Darolutamide in Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Abemaciclib Plus Darolutamide in Prostate Cancer That Has Spread After Initial Treatment
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18714; I3Y-MC-JPEI (Other: Eli Lilly and Company); 2023-503919-15-00 (Other: EU Trial Number); U1111-1294-1466 (Registry Identifier: WHO Universal Trial Number (UTN))
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abemaciclib; darolutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib + Darolutamide (Experimental): Abemaciclib plus (+) darolutamide. Participants who have not undergone bilateral orchiectomy are required to continue background androgen deprivation therapy (ADT) with a luteinizing hormone-releasing hormone (LHRH) agonist/antagonist throughout the study.
  Interventions: Drug: Abemaciclib; Drug: Darolutamide; Drug: LHRH agonist/antagonist

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219
Drug: Darolutamide — Administered orally.
Drug: LHRH agonist/antagonist — Physician's choice. Administered in accordance with the prescribing information.

SUMMARY:
The main purpose of this study is to learn more about the safety and tolerability of abemaciclib when given in combination with darolutamide to participants with prostate cancer that has spread after initial treatment. Participation may last up to 32 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Metastatic castration-resistant prostate cancer evidenced by:

  * Prostate-specific antigen (PSA) or radiographic progression despite castrate levels of testosterone
  * At least 1 bone metastasis on bone scan and/or 1 soft tissue metastasis on computed tomography/magnetic resonance imaging (CT/MRI)
* Participants who have not undergone bilateral orchiectomy must continue luteinizing-hormone-releasing hormone (LHRH) agonists/antagonists throughout the study.
* Have adequate organ function.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.

Exclusion Criteria:

* Prior treatment with cyclin-dependent kinase 4 and 6 (CDK4 and CDK6) inhibitors or darolutamide.
* Prior systemic therapy for metastatic castration-resistant prostate cancer(mCRPC) with cytotoxic chemotherapy, PARP inhibitors, novel hormonal agents (NHAs) (enzalutamide, apalutamide, and abiraterone), and radiopharmaceuticals.
* Serious preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
* Clinically significant heart disease as evidenced by myocardial infarction, arterial thrombotic events, severe or unstable angina, or congestive heart failure (New York Heart Association Class III or IV) within 6 months of assignment to treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Date of first dose to study completion (approximately 32 months)
  Administration Number of Participants with One or More SAEs Considered by the Investigator to be Related to Study Drug Administration

SECONDARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) Assessed by Investigator rPFS Assessed by Investigator | Date of first dose to radiographic disease progression or death from any cause (approximately 32 months)
  rPFS Assessed by Investigator
Objective Response Rate (ORR): Percentage of Participants with Soft Tissue Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) | Date of first dose to radiographic disease progression or death from any cause (approximately 32 months)
  ORR: Percentage of Participants with Soft Tissue BOR of CR or PR
Duration of Response (DoR) | Date of first documented CR or PR to radiographic disease progression or death from any cause (approximately 32 months)
  DOR
Time to Prostate Specific Antigen (PSA) Progression | Date of first dose to the first observation of PSA progression (approximately 32 months)
  Time to PSA progression
Prostate Specific Antigen (PSA) Response Rate (PSA-RR): Percentage of Participants with a PSA Decrease of at Least 50% from Baseline | Date of first dose to confirmed PSA progression (approximately 32 months)
  PSA-RR
Pharmacokinetics (PK): Mean Concentrations of Abemaciclib and its Active Metabolite(s) | Cycle 1 Day 1 until Cycle 2 Day 1 (Cycle = 28 days)
  PK: Mean Concentrations of Abemaciclib and its Active Metabolite(s)
Pharmacokinetics (PK): Mean Concentrations of Darolutamide and its Active Metabolite | Cycle 1 Day 1 until Cycle 2 Day 1 (Cycle = 28 days)
  PK: Mean Concentrations of Darolutamide and its Active Metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (3):
  - Highlands Oncology Group, Springdale, Arkansas
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
- Germany (4):
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Klinikum Rechts Der Isar Der Technischen Universität München, Munich, Bavaria
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Spain (6):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Abemaciclib Plus Darolutamide in Prostate Cancer That Has Spread After Initial Treatment — https://trials.lilly.com/en-US/trial/418175